CLINICAL TRIAL: NCT07329283
Title: Nighttime Synchrony of Your Nutrition and Circadian Health: The N-Sync Study
Brief Title: Nighttime Synchrony of Your Nutrition and Circadian Health
Acronym: N-Sync
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Depner, PhD, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 185590
Record Dates: First submitted 2025-12-11; First posted 2026-01-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sleep; Metabolism Changes; Circadian Rhythm; Lifestyle Factors; Sleep Hygiene; Sleep Hygiene, Inadequate; Sleep Deprivation; Insufficient Sleep; Circadian Misalignment; Circadian Dysregulation; Light Exposure
Keywords: Sleep; Light Exposure; Metabolism; Circadian Rhythm; Food Intake; Lifestyle Factors; Sleep Hygiene
MeSH Terms: conditions — Sleep Hygiene; Sleep Deprivation; Chronobiology Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization to condition order will be concealed to research staff and participants until the conclusion of the condition "A", which all participants will complete first.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sleep Restriction with Central and Peripheral Alignment (No Intervention): (Arm "A")-Control condition with central and peripheral aligned circadian rhythms
- Sleep Restriction with Central Clock Misalignment (Experimental): (Arm "B")-Misalignment of the central clock by nighttime electrical light exposure and dim-light in morning hours.
  Interventions: Behavioral: Central Clock Misalignment
- Sleep Restriction with Peripheral Misalignment (Experimental): (Arm "C")-Misalignment of peripheral oscillators by shifting the majority of food intake to the nighttime hours.
  Interventions: Behavioral: Peripheral Misalignment

INTERVENTIONS:
Behavioral: Central Clock Misalignment — Light exposure will be dimmed during the first 4 hours of scheduled wakefulness, with bright light exposure during the nighttime hours of extended wakefulness.
  Arms: Sleep Restriction with Central Clock Misalignment
Behavioral: Peripheral Misalignment — Most daily calories will be given later in the day to shift eating patterns toward the nighttime hours.
  Arms: Sleep Restriction with Peripheral Misalignment

SUMMARY:
Sleep is an important factor for overall health. This study will see how different light exposure patterns and food intake impact a person's metabolism (how the body breaks down food) when sleeping is reduced.

Participants will attend 6 to 8 in-person visits to the study clinic, including three overnight stays. People will complete surveys and medical tests. The study will last about 4 to 6 months.

DETAILED DESCRIPTION:
This study is a randomized in-lab, cross-over trial. Each participant will complete all three arms in either condition order #1 (A-B-C) or order #2 (A-C-B). Each arm will consist of 5 nights of experimental sleep restriction followed by a constant routine protocol for assessment of 24-h rhythms. Sleep restriction in the three arms will occur under the following conditions: (A-control condition) Sleep Restriction with Central and Peripheral Alignment; (B) Sleep Restriction with Central Clock Misalignment; and (C) Sleep Restriction with Peripheral Misalignment. Prior to enrollment participants will complete a comprehensive medical history and clinical overnight sleep disorders screening. Baseline consists of a ~2-week ambulatory real-world monitoring segment that will occur immediately prior to each in-lab sleep restriction condition. Following the 5 days of sleep restriction in each arm, participants will complete an intravenous glucose tolerance test to analyze insulin sensitivity, prior to completing the constant routine.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-35 years old; equal numbers of men and women
2. Body Mass Index (BMI): 18.5-24.9 kg/m2
3. Sleep Habits: habitual self-reported average total sleep time (TST) 7-9 hours per night for prior 6 months

Exclusion Criteria:

1. Clinically diagnosed sleep disorder or apnea hypopnea index (AHI) ≥5
2. Evidence of significant organ system dysfunction or disease (e.g., heart disease, diabetes)
3. Fasting plasma glucose ≥100 mg/dL
4. Major psychiatric illness (e.g., major depressive disorder)
5. Cancer that has been in remission less than 5 years
6. History of shift-work in prior year
7. Weight change >5% of body weight over prior six months
8. Currently following a weight-loss program
9. Menopause
10. Pregnant/nursing
11. Greater than 5-day variation in menstrual cycle length month-to-month
12. Currently smoking
13. Alcohol intake >14 drinks/week or >3 drinks/day.
14. Use of prescription medications (except oral contraceptives) within one month prior to or during in-lab visits.
15. Consumption of illegal drugs or >500mg per day of caffeine.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | Immediately following the 5-day sleep restriction segment
  Insulin sensitivity will be measured by intravenous glucose tolerance tests.
Internal Circadian Misalignment (Uridine and Isobutyryl-L-carnitine) | During the constant routine, following the 5-day sleep restriction segment
  Phase angle between DLMO and acrophase of uridine and isobutyryl-L-carnitine during constant routine.

OTHER OUTCOMES:
Timing of DLMO and DLMOff | During the constant routine, following the 5-day sleep restriction segment
  The phase angle between dim-light melatonin offset (DLMOff) scheduled waketime using hourly saliva samples collected during a constant routine.
Hunger and Satiety Visual Analog Scales | During the constant routine, following the 5-day sleep restriction segment
  Self-reported ratings of hunger, satiety, and prospective food intake will be quantified by 100mm visual analog scales ranging from 0 to 100. For each scale, 0 represents low hunger, satiety, or prospective food intake, with 100 representing the highest hunger, satiety, or prospective food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Depner, PhD, Principal Investigator — University of Utah
Locations (1):
- College of Health Research Complex - University of Utah, Salt Lake City 84112, Salt Lake City, Utah, United States